CLINICAL TRIAL: NCT03901313
Title: A Phase 1, Open-Label, Randomized, 3-Period Crossover Study to Assess the Effect of Low-Fat Food on Pexidartinib Pharmacokinetics in Healthy Subjects
Brief Title: Effect of Low-Fat Food on Pexidartinib Pharmacokinetics in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: PL3397-A-U128
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Results first posted 2020-04-22 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-04

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics
MeSH Terms: interventions — pexidartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Sequence ABC (Experimental): Healthy volunteers will receive Treatments A, then B, and then C, with a 6-day washout between treatments, during a stay at the clinic of 20 days
  Interventions: Drug: Treatment A - 400 mg Fasting; Drug: Treatment B - 400 mg Fed; Drug: Treatment C - 200 mg Fed
- Sequence ACB (Experimental): Healthy volunteers will receive Treatments A, then C, and then B, with a 6-day washout between treatments, during a stay at the clinic of 20 days
  Interventions: Drug: Treatment A - 400 mg Fasting; Drug: Treatment B - 400 mg Fed; Drug: Treatment C - 200 mg Fed
- Sequence BAC (Experimental): Healthy volunteers will receive Treatments B, then A, and then C, with a 6-day washout between treatments, during a stay at the clinic of 20 days
  Interventions: Drug: Treatment A - 400 mg Fasting; Drug: Treatment B - 400 mg Fed; Drug: Treatment C - 200 mg Fed
- Sequence BCA (Experimental): Healthy volunteers will receive Treatments B, then C, and then A, with a 6-day washout between treatments, during a stay at the clinic of 20 days
  Interventions: Drug: Treatment A - 400 mg Fasting; Drug: Treatment B - 400 mg Fed; Drug: Treatment C - 200 mg Fed
- Sequence CAB (Experimental): Healthy volunteers will receive Treatments C, then A, and then B, with a 6-day washout between treatments, during a stay at the clinic of 20 days
  Interventions: Drug: Treatment A - 400 mg Fasting; Drug: Treatment B - 400 mg Fed; Drug: Treatment C - 200 mg Fed
- Sequence CBA (Experimental): Healthy volunteers will receive Treatments C, then B, and then A, with a 6-day washout between treatments, during a stay at the clinic of 20 days
  Interventions: Drug: Treatment A - 400 mg Fasting; Drug: Treatment B - 400 mg Fed; Drug: Treatment C - 200 mg Fed

INTERVENTIONS:
Drug: Treatment A - 400 mg Fasting — Single oral 400 mg (2 × 200 mg capsules) dose of pexidartinib in the morning under fasting conditions
  Other Names: Pexidartinib
Drug: Treatment B - 400 mg Fed — Single oral 400 mg (2 × 200 mg capsules) dose of pexidartinib in the morning within 30 minutes (min) after a low-fat standard breakfast meal
  Other Names: Pexidartinib
Drug: Treatment C - 200 mg Fed — Single oral 200 mg (1 × 200 mg capsule) dose of pexidartinib in the morning within 30 min after a low-fat standard breakfast meal
  Other Names: Pexidartinib

SUMMARY:
All participants in this study are healthy volunteers.

Throughout the study, healthy volunteers will have physical exams, electrocardiograms and clinical laboratory tests. The study staff will keep track of symptoms, diet, and what medications they are taking.

Each participant will get all three treatments (A, B and C). Only the order in which they receive them will be different.

There are six groups based on the order: ABC, ACB, BAC, BCA, CAB, or CBA. Participants have an equal chance of being assigned to any of these groups.

For each treatment period, participants will:

* fast overnight
* receive the assigned treatment with or without food
* have a small tube of blood drawn prior to treatment
* after dosing, additional blood samples will be drawn at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 14, 22, 24, 28, 32, 36, 48, 54, 60, 72, 84, 96, 108, 120, 132, and 144 hours
* have a break from treatment for 6 days between each treatment period

All participants must reside in the clinic for a total of 20 days.

DETAILED DESCRIPTION:
The primary objectives of this study are:

* To assess the effect of low-fat food on the pharmacokinetics (PK) of pexidartinib following a single oral dose of 400 mg administered in healthy subjects
* To assess the PK of pexidartinib following a single oral dose of 200 mg administered with low-fat food in healthy subjects

The secondary objective of this study is:

* To characterize the safety and tolerability of pexidartinib in healthy subjects following administration of a single oral dose of pexidartinib with low fat food and without food

ELIGIBILITY:
Inclusion Criteria:

* Is healthy at screening visit
* Is not pregnant or lactating
* Is surgically or naturally unable to reproduce, or agrees to remain sexually abstinent or to use double barrier methods of contraception from check-in until 90 days after the final dose of pexidartinib
* Has a Body Mass Index (BMI) of 18-30 kg/m^2, inclusive
* Has negative test results for protocol-defined drugs and diseases at screening and/or check-in
* Is willing to avoid food or beverages before check-in until the end of the study:

  1. containing caffeine/xanthine or alcohol from 48 hours before check-in
  2. containing grapefruit or Seville oranges 6 days before check-in

Exclusion Criteria:

* Per protocol or in the opinion of the investigator at screening and/or check-in, has something that would preclude participation:

  1. has a clinically significant disorder, disease or lab value
  2. consumes a prohibited drug, drink or food
  3. is unable to consume the standard meal
* Is an employee of the clinic or their family member

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-05-08 (Actual); Study Completion 2019-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 24 participants who met all inclusion criteria and no exclusion criteria were enrolled in the study.
Period: Overall Study
Arm/Group | Sequence ABC | Sequence ACB | Sequence BAC | Sequence BCA | Sequence CAB | Sequence CBA
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Healthy volunteers randomized to receive 1 of 6 sequences of Treatment A, B, and C, with a 6-day washout between treatments, during a stay at the clinic of 20 days
  Treatment A - 400 mg Fasting: Single oral 400 mg (2 × 200 mg capsules) dose of pexidartinib in the morning under fasting conditions
  Treatment B - 400 mg Fed: Single oral 400 mg (2 × 200 mg capsules) dose of pexidartinib in the morning within 30 minutes (min) after a low-fat standard breakfast meal
  Treatment C - 200 mg Fed: Single oral 200 mg (1 × 200 mg capsule) dose of pexidartinib in the morning within 30 min after a low-fat standard breakfast meal
Arm/Group | All Participants
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.6 (8.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Concentration in Plasma (Cmax) of Pexidartinib
Description: Mean Cmax of pexidartinib is calculated for each treatment period
Time Frame: Baseline, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 14, 22, 24, 28, 32, 36, 48, 54, 60, 72, 84, 96, 108, 120, 132, and 144 hours postdose
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Treatment A: All healthy volunteers who received Treatment A - 400 mg Fasting: Single oral 400 mg (2 × 200 mg capsules) dose of pexidartinib in the morning under fasting conditions
- Treatment B: All healthy volunteers who received Treatment B - 400 mg Fed: Single oral 400 mg (2 × 200 mg capsules) dose of pexidartinib in the morning within 30 minutes (min) after a low-fat standard breakfast meal
- Treatment C: All healthy volunteers who received Treatment C - 200 mg Fed: Single oral 200 mg (1 × 200 mg capsule) dose of pexidartinib in the morning within 30 min after a low-fat standard breakfast meal
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 24 | 24 | 24
ng/mL | 4580 (1240) | 7090 (1590) | 3870 (729)

2. Primary Outcome: Time to Cmax (Tmax)
Description: Median Tmax of pexidartinib is calculated for each treatment period
Time Frame: as for outcome 1
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Median (Full Range); unit: hours
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 24 | 24 | 24
hours | 2.00 [1.00 to 3.52] | 3.50 [2.50 to 10.00] | 3.30 [2.50 to 4.50]

3. Primary Outcome: Area Under the Concentration-time Curve From Time of Dosing to Last Measurable Concentration (AUClast) and to Infinity (AUCinf)
Description: Mean AUClast and AUCinf for pexidartinib are calculated for each treatment period
Time Frame: as for outcome 1
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng*hour/mL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 24 | 24 | 24
ng*hour/mL
  AUClast | 64800 (19300) | 102000 (26300) | 53600 (14200)
  AUCinf | 66100 (19900) | 104000 (27400) | 54600 (15000)

4. Primary Outcome: Terminal Half-life (t1/2)
Description: Mean t1/2 for pexidartinib is calculated for each treatment period
Time Frame: as for outcome 1
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 24 | 24 | 24
hours | 24.2 (5.28) | 23.1 (4.68) | 23.6 (5.04)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from study enrollment up to 28 days of administration of the last dose of study treatment.
Description: A treatment-emergent adverse event (TEAE) was defined as an adverse event that emerged during treatment, having been absent pre-treatment, or worsened relative to the pre-treatment state.
Arm/Group | Treatment A | Treatment B | Treatment C
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 1/24 | 0/24 | 2/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=24) | Treatment B (N=24) | Treatment C (N=24)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/13/NCT03901313/Prot_SAP_000.pdf